CLINICAL TRIAL: NCT04277364
Title: Effects of Phosphatidic Acid Supplementation on Strength and Hypertrophic Responses to Strength Training
Brief Title: Effects of Phosphatidic Acid on Strength and Hypertrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA strength adaptations
Record Dates: First submitted 2020-02-09; First posted 2020-02-20 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Hypertrophy; Muscle Strength
Keywords: Dietary Supplementations; Athletic Performance; Phosphatidic acid
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- High dose phosphatidic acid (Active Comparator): 750mg of phosphatidic acid per day for 8 weeks
  Interventions: Dietary Supplement: phosphatidic acid supplementation; Other: Strength training
- Low dose phosphatidic acid (Active Comparator): 375mg of phosphatidic acid per day for 8 weeks
  Interventions: Dietary Supplement: phosphatidic acid supplementation; Other: Strength training
- Placebo (Placebo Comparator): 750mg of corn starch per day for 8 weeks
  Interventions: Other: Placebo (corn starch supplementation); Other: Strength training

INTERVENTIONS:
Dietary Supplement: phosphatidic acid supplementation — The total daily doses will be distributed in 3 individual doses: in the group that will ingest 750mg per day, the individual doses will be 250mg, while in the group that will ingest 375mg per day, the individual doses will be 125mg. The capsules should be consumed at breakfast, 30 minutes before each training session (or at lunch, on days when there is no training) and at dinner.
  Arms: High dose phosphatidic acid; Low dose phosphatidic acid
Other: Placebo (corn starch supplementation) — Three individual doses of corn starch will be consumed per day. The capsules should be consumed at breakfast, 30 minutes before each training session (or at lunch, on days when there is no training) and at dinner.
  Arms: Placebo
Other: Strength training — All participants will be submitted to a 8-week strength training program, with 3 training sessions per week, totaling 24 training sessions.

SUMMARY:
There are indications that phosphatidic acid (PA) supplementation is capable of enhancing gains in strength and muscle mass in response to strength training, although the literature is still incipient and controversial. Given the possible benefits in terms of maintenance and increased skeletal muscle mass, which still need confirmation, this study aims to examine the effectiveness of PA supplementation in two different doses in increasing skeletal muscle mass and strength in adult men undergoing to 8 weeks of strength training. For this, about 45 men will be randomly allocated to one of three treatments at a ratio of 1:1:1: PA 750mg per day, PA 375mg per day, or placebo (cornstarch, 750mg per day). All participants will undergo a 8-week strength training program, 3 times a week, totaling 24 sessions, which will begin with the start of supplementation. Individuals will be assessed for maximum dynamic strength of upper and lower limbs, resistance to dynamic strength of upper and lower limbs, body composition, muscle cross-sectional area and food consumption. Samples of venous blood will also be collected to determine the concentration of creatine kinase (CK), lactate dehydrogenase (LDH), testosterone, insulin-like growth factor type 1 (IGF-1), growth hormone (GH) and cortisol. These evaluations will be carried out before (PRE) and after (POST) the period of supplementation and training. Additional blood samples will be taken 48 hours after the first and last training sessions, for specific determination of blood muscle damage markers: CK and LDH.

DETAILED DESCRIPTION:
There are indications that phosphatidic acid (PA) supplementation is capable of enhancing gains in strength and muscle mass in response to strength training, although the literature is still incipient and controversial. The present study will adopt a randomized, double-blind, parallel group and placebo-controlled design, with the objective of evaluating the effectiveness of chronic phosphatidic acid supplementation in gaining maximum dynamic muscle strength, body composition and muscle cross-sectional area in trained adult individuals submitted to a strength training program.

About 45 men will be randomly allocated to one of the three treatments, in the proportion 1: 1: 1: PA 750mg per day, PA 375 per day, or placebo (corn starch, 750 per day), for 8 weeks. The allocation of participants to the experimental groups will be randomized using software (www.random.org). In addition to the pairing, the groups will be equalized by the maximum dynamic force (sum of the upper and lower limb loads) of the participants at the PRE moment. For randomization, proportional distribution between groups and equalization by maximum force, participants will be recruited in blocks of 6 or 9 participants, which will be ranked based on their maximum strength, with these procedures being carried out within each block. Random sequences of numbers 1, 2 and 3, representing the treatments PA high dose, PA low dose and placebo, will be randomly distributed to each three participants within each block, respecting the ranking by maximum force.

All participants will be submitted to a 8-week strength training program, 3 times a week, totaling 24 sessions, which will start at the beginning of supplementation. The training will follow the daily wavy periodization model.In this model, the weekly training sessions are called A, B and C, with the total volume changed at each session, as follows: in sessions A, participants will do 3 sets of each exercise, in sessions B, 4 sets of each exercise and, in sessions C, again 3 sets of each exercise. Participants will perform the following exercises: bench press, 45º leg-press, pulley pull, squat on the guided bar and leg extension in the extension chair. The interval between sets will be 60 seconds and, between exercises, 90 seconds. The loads will be individually adjusted for each series, in such a way that the participants are able to perform between 8 and 12 maximum repetitions (until the concentric failure or until the participant cannot maintain an adequate pattern of movement).

Before and after treatments, participants will be evaluated for the following parameters: body composition, maximum dynamic strength of upper limbs (1RM supine) and lower limbs (1RM leg-press), dynamic strength resistance of upper and lower limbs, cross-sectional area of the vastus lateralis and rectus femoris muscles via ultrasound.The following blood parameters will also be evaluated: CK, LDH, free testosterone, IGF-1, GH and cortisol through immunoenzymatic, colorimetric enzymatic or fluorimetric enzymatic assays. Additional blood collections will be performed 48 hours after the first and last sessions training for specific determination of blood muscle damage markers: CK and LDH.

The assessment of maximum strength will be performed on leg-press equipment, for the lower limbs, and supine, for the upper limbs. The tests for assessing maximum dynamic strength (1RM) will follow methods proposed by the American Society for Exercise Physiology (Brown & Weir, 2001). The evaluation of dynamic strength endurance will be performed in leg-press and bench press exercises where the volunteers must perform repetitions until fatigue with a load equivalent to 70% of 1RM, which will be previously determined in the maximum strength test. Participants will have to perform the maximum number of repetitions until reaching the concentric failure. Each individual will perform 3 sets with an interval of 2 minutes between them.

Body composition will be assessed by dual emission densitometry with X-ray source (DXA), using the Hologic QDR 4500 Discovery Densitometer (Hologic Inc., Bedford, MA, USA).

The architecture of the vastus lateralis and rectus femoris muscles will be evaluated with a B-mode ultrasound, with a linear vector transducer and a frequency of 7.5 MHz (Samsung, Sonaance R3). The images obtained will be assembled in such a way that the cross-sectional area of the vast side is established, which will be subsequently evaluated by the Madena 3.2.1 free-use image digitization software.

The evaluation of food consumption will be carried out through food diaries of 3 non-consecutive days, two of which are weekdays, and one weekend. Energy and macronutrient consumption will be calculated using the Nutritionist Pro software.

The data obtained in the PRE-intervention period will be compared between the groups using one-way ANOVA after confirmation of the normality of the data distribution, which will be done using the Shapiro-Wilk test. If the distribution is not normal, the Kruskal-Wallis non-parametric test will be used. All study variables will be evaluated following the mixed 2-factor model (time and group), with two levels in the time factor (PRE vs. POST) and three levels in the treatment factor (high dose vs. low dose BP vs. Placebo). Participants will be random factors. Four different covariance matrix structures will be tested and the one that demonstrates the best fit to each data set will be used (lowest BIC, or Bayes information criterion). If there is a statistically significant interaction effect, a hypothesis-guided contrast analysis of degree of freedom will be conducted to locate intra- and inter-subject differences.

Post-pre deltas will also be calculated, both in percentage and absolute terms, for all variables. These data will be compared between groups by means of one-way ANOVA, or by Kruskal-Wallis test, if they do not present a normal distribution. The data will be presented in mean and standard deviation. The analyzes will be made using the SAS 9.3 software. The level of significance adopted will be 5%.

The sample size was determined with the aid of the G-Power software (v. 3.1.9.2) considering the F test model (ANOVA with repeated measures), with comparisons within and between, with three groups being evaluated twice in time. The input parameters were: significance level = 5%; effect size = 0.25 (small); power (1-β) = 0.8, which resulted in a total sample size of 42 participants. To account for probable sample losses and dropouts, around 45 participants will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* 6 months of continuous strength training, with a minimum weekly volume of 3 hours of training
* Minimum dynamic maximum strength index of 1.1 times the body weight for bench press and 2.5 times the body weight for leg press
* Consume> 1.7g of protein per kilo of body weight in their diets
* Keeping body weight stable in the 3 months prior to the study

Exclusion Criteria:

* History of use of anabolic-androgenic steroids
* Smoking
* Use of dietary supplements that may affect strength or muscle mass in the last 3 months before the study
* Presence of infectious disease in the last 4 weeks prior to the study
* Chronic use of drugs that can potentially affect the variables that will be assessed
* Any condition that prevents the performance of maximum strength tests or strength training

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare muscle strength responses | 8 weeks
  Assessments of the maximum dynamic strength and the dynamic strength resistance of the upper and lower limbs will be performed before and after treatment. The evaluation of the maximum dynamic strength will be performed on leg-press equipment, for the lower limbs, and bench press, for the upper limbs. The tests for assessing maximum dynamic strength (1RM) will follow methods proposed by the American Society for Exercise Physiology (Brown & Weir, 2001). After determining the 1-RM, the test will be repeated 5 days later to confirm the maximum loads. The tests will be repeated as many times as necessary until the difference between charges is less than 5%. The evaluation of dynamic strength endurance will be performed in leg-press and bench press exercises where the volunteers must perform repetitions until fatigue with a load equivalent to 70% of 1RM. Participants will have to perform the maximum number of repetitions until reaching the concentric failure.
Compare muscle hypertrophy responses | 8 weeks
  The architecture of the vastus lateralis and rectus femoris muscles will be evaluated with a B-mode ultrasound, with a linear vector transducer and a frequency of 7.5 MHz (Samsung, Sonaance R3).For this, the volunteers will be placed in the supine position with legs extended. An experienced researcher will delimit, with semi-permanent ink, the point on which the measurements will be taken. The skin will then be marked transversely (angle of 90 with the lateral epicondyle of the tibia) every 2 cm for measurements. The transducer, aligned perpendicular to the muscle, will be moved from a central position to a lateral position along the pre-established boundaries. The contact pressure will be kept minimal and stable during each measurement. Finally, the images obtained will be assembled in such a way that the cross-sectional area of the vast side is established, which will be subsequently evaluated by the Madena 3.2.1 free-use image digitization software.

SECONDARY OUTCOMES:
Assess effects on body composition | 8 weeks
  Body composition will be assessed by dual emission densitometry with X-ray source (DXA), using the Hologic QDR 4500 Discovery Densitometer (Hologic Inc., Bedford, MA, USA). For the assessment of body composition using the DXA device, the participant will have to lie down in the supine position, remaining at rest during the exam. All assessments will be carried out by a qualified technician with previous protocol experience.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Giannini Artioli, phD, Study Chair — School of Physical Education and Sport, University of São Paulo
Locations (1):
- School of Physical Education and Sports, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No